CLINICAL TRIAL: NCT04075201
Title: A Phase ⅠClinical Trial of Recombinant Hepatitis B Vaccine (Hansenula Polymorpha, 10μg) With an Open-labelled Design in Adults and a Randomized, Double-blinded, Positive Controlled Design in Children and Neonates
Brief Title: Clinical Trial of Recombinant Hepatitis B Vaccine (Hansenula Polymorpha, 10μg)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO-HB-1001
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: Single group in the adults participants, and parallel groups in the children and neonates participants.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Open-labelled in the adults participants, and double-blinded in the children ans neonates participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Adults-Experimental group (Experimental): One dose of investigational vaccine
  Interventions: Biological: One dose of investigational vaccine
- Children-Experimental group (Experimental): One dose of investigational vaccine
  Interventions: Biological: One dose of investigational vaccine
- Children-Control group (Active Comparator): One dose of control vaccine
  Interventions: Biological: One dose of control vaccine
- Neonates-Experimenatal group (Experimental): Three doses of investigational vaccine
  Interventions: Biological: Three doses of investigational vaccine
- Neonates-Control group (Active Comparator): Three doses of control vaccine
  Interventions: Biological: Three doses of control vaccine

INTERVENTIONS:
Biological: One dose of investigational vaccine — One dose of investigational hepatitis B vaccine (10μg/0.5ml) developed by Sinovac Research & Development Co., Ltd.
  Arms: Adults-Experimental group; Children-Experimental group
Biological: One dose of control vaccine — One dose of control hepatitis B vaccine (10μg/0.5ml) manufactured by Dalian Hissen Bio-pharmInc.
  Arms: Children-Control group
Biological: Three doses of investigational vaccine — Three doses of investigational hepatitis B vaccine (10μg/0.5ml) developed by Sinovac Research & Development Co., Ltd. on the schedule of month 0,1,2
  Arms: Neonates-Experimenatal group
Biological: Three doses of control vaccine — Three doses of control hepatitis B vaccine (10μg/0.5ml) manufactured by Dalian Hissen Bio-pharmInc.
  Arms: Neonates-Control group

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of the recombinant hepatitis B vaccine (Hansenula polymorpha, 10μg), with an open-labelled design in adults and randomized, double-blinded, and positive controlled design in children and neonates.

DETAILED DESCRIPTION:
This is a phase Ⅰ clinical trial of recombinant hepatitis B vaccine (Hansenula polymorpha,10μg) with an open-labelled design in adults and randomized, double-blinded, and positive controlled design in children and neonates. The control vaccine was the commercialized recombinant hepatitis B vaccine (Hansenula polymorpha,10μg) manufactured by Dalian Hissen Bio-pharm Lnc. Twenty four adults aged from 18 to 49 years will be vaccinated with one dose of investigational vaccine. Sixty children aged from 1 to 15 years will be randomly assigned in a 1:1 ratio to receive one dose of in investigational vaccine or control vaccine. Sixty neonates will be randomly assigned in a 1:1 ratio to receive three doses of investigational vaccine or control vaccine on the schedule of month 0,1,2. Safety profiles 30 days after each dose will be assessed based on all the participants, and immunogenicity will be assessed based on the enrolled chidren and neonates.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18~49 years, or children aged 1~15 years, or neonates within 24 hours of birth;
* Proven legal identity;
* Participants or guardians of the participants should be capable of understanding the written consent form, and such form should be signed prior to enrollment ;

Exclusion Criteria (For Adults):

* Breast feeding, pregnant, or expected to conceive in the next 60 days;
* History of allergy to any vaccine or vaccine ingredient, or serious adverse reaction(s) to vaccination, such as urticaria, difficulty in breathing, angioneurotic edema, abdominal pain, etc;
* Congenital malformation, developmental disorders, genetic defects;
* Autoimmune disease or immunodeficiency/immunosuppressive;
* Severe chronic diseases, severe cardiovascular disease, hypertension and diabetes that cannot be controlled by drugs, liver Kidney disease, malignant tumor;
* Severe nervous system disease or mental illness;
* Asplenia or functional asplenia;
* Diagnosed coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities) , or obvious bruising or coagulation disorders;
* Any immunosuppressant, cytotoxic medicine, or inhaled corticosteroids (except corticosteroid spray for treatment of allergic rhinitis or corticosteroid treatment on surface for acute non-complicated dermatitis) within 6 month prior to study entry;
* Long term history of alcoholism or drug abuse;
* Administration of blood product within 3 months prior to the entry;
* Administration of any other investigational drugs within 30 days prior to the entry;
* Receipt of any attenuated live vaccine within 14 days prior to study entry;
* Receipt of any subunit vaccine or inactivated vaccine within 7 days prior to study entry;
* Any acute disease within 7 days prior to the study entry;
* Axillaty temperature > 37.0 °C;
* Any other factor that suggesting the volunteer is unsuitable for this study based on the opinions of investigators.

Exclusion Criteria (For Children):

* History of extra vaccination of Hepatitis B vaccine or vaccine containing hepatitis B except for the primary vaccination in the immunization planning program;
* History of allergy to any vaccine or vaccine ingredient, or serious adverse reaction(s) to vaccination, such as urticaria, difficulty in breathing, angioneurotic edema, abdominal pain, etc;
* Congenital malformation, developmental disorders, genetic defects;
* Autoimmune disease or immunodeficiency/immunosuppressive;
* Severe chronic diseases, severe cardiovascular disease, hypertension and diabetes that cannot be controlled by drugs, liver Kidney disease, malignant tumor;
* Severe nervous system disease or mental illness;
* Asplenia or functional asplenia;
* Diagnosed coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities) , or obvious bruising or coagulation disorders;
* Any immunosuppressant, cytotoxic medicine, or inhaled corticosteroids (except corticosteroid spray for treatment of allergic rhinitis or corticosteroid treatment on surface for acute non-complicated dermatitis) within 6 month prior to study entry; Long term history of alcoholism or drug abuse;
* Administration of blood product within 3 months prior to the entry;
* Administration of any other investigational drugs within 30 days prior to the entry;
* Receipt of any attenuated live vaccine within 14 days prior to study entry;
* Receipt of any subunit vaccine or inactivated vaccine within 7 days prior to study entry;
* Any acute disease within 7 days prior to the study entry;
* Axillaty temperature > 37.0 °C;
* Any other factor that suggesting the volunteer is unsuitable for this study based on the opinions of investigators.

Exclusion Criteria (For Neonates):

* Neonates gestational age <37 weeks or >42 weeks;
* Birth weight <2500g for boy, <2300g for girl;
* Apgar score at birth <8;
* Positive for any of the mother's HBsAg, HBeAg, HBeAb, and HBcAb (check the laboratory report of the birth hospital);
* Parents have family history of convulsions, epilepsy, encephalopathy, etc.;
* Mother's immune function is low or history of organ transplantation or hemodialysis;
* Mother has history of allergy to any vaccine or vaccine ingredient, or serious adverse reaction(s) to vaccination, such as urticaria, difficulty in breathing, angioneurotic edema, abdominal pain, etc;
* Family history of coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities) , or obvious bruising or coagulation disorders;
* Immune system function damage, or parents have autoimmune diseases or immunodeficiency/immunosuppression;
* Congenital malformation, developmental disorders, genetic defects;
* Diognosed or suspected of active infection, cardiovascular disease, etc.;
* Axillaty temperature > 37.0 °C;
* Any other factor that suggesting the volunteer is unsuitable for this study based on the opinions of investigators.

Max Age: 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2019-07-07 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-07-25 (Actual)

PRIMARY OUTCOMES:
The overall incidence of the adverse reactions after each dose vaccination | within 30 days after each dose
  Safety index-After each dose, a 30-minute safety observation will be conducted immediately. The body temperature, solicited local and general adverse events (AE) on day 0-7 were reported. The solicited local symptoms include pain, induration, redness, swelling, rash, and pruritus. The solicited general adverse symptoms include allergy, fatigue, irritability, inappetence, vomiting, diarrhea, and fever. Unsolicited adverse events on day 0-30 were also reported, which include the unsolicited symptoms happened within 0-7 days, and any symptoms happened within the 8-28 days. Each AE case will be reviewed by the investigator to determine whether it was an adverse reaction (The vaccination-related AE). The incidence of adverse reactions=Number of subjects who have adverse reactions of any symptoms/number of all the subjects whose safety information are collected.

SECONDARY OUTCOMES:
The incidence of the serious adverse events (SAEs) | For adults and children: 30 days; for neonates: 18 months
  Safety index-After each dose, the serious adverse events in the safety observation period will be reported.
  The SAE incidence=Number of subjects who have SAE of any symptoms/Number of subjects whose safety information are collected.
The seroconversion rate (SCR) of anti-HBs 1 months after the single dose injection in Children aged 1-15 years | 30 days after the injection
  Immunogenicity index-Subjects whose pre-immune anti-HBs concentration <10mIU/ml, and post-immune anti-HBs concentration ≥10mIU/ml, or those whose pre-immune anti-HBs concentration ≥10mIU/ml and the increase of post-immune anti-HBs level ≥4 folds are considered seroconverted.
The geometric mean concentration (GMC) of anti-HBs 1 months after the single dose injection in Children aged 1-15 years | 30 days after the injection
  Immunogenicity index
The SCR of anti-HBs 7 months after the first dose injection in neonates | 210 days after the first dose injection
  Immunogenicity index-Subjects whose pre-immune anti-HBs concentration <10mIU/ml, and post-immune anti-HBs concentration ≥10mIU/ml, or those whose pre-immune anti-HBs concentration ≥10mIU/ml and the increase of post-immune anti-HBs level ≥4 folds are considered seroconverted.
The GMC of anti-HBs 7 months after the first dose injection in neonates | 210 days after the first dose injection
  Immunogenicity index
The SCR of anti-HBs 2 months after the first dose injection in neonates | 60 days after the first dose injection
  Immunogenicity index-Subjects whose pre-immune anti-HBs concentration <10mIU/ml, and post-immune anti-HBs concentration ≥10mIU/ml, or those whose pre-immune anti-HBs concentration ≥10mIU/ml and the increase of post-immune anti-HBs level ≥4 folds are considered seroconverted.
The GMC of anti-HBs 7 months after the first dose injection in neonates | 60 days after the first dose injection
  Immunogenicity index

CONTACTS AND LOCATIONS:
Overall Officials: Shengli Xia, Doctor, Principal Investigator — Henan Provincial Center for Disease Control and Prevention
Locations (1):
- Biyang County Center for Disease Control and Prevention, Zhumadian, Henan, China